CLINICAL TRIAL: NCT02472301
Title: Randomized, Single-blinded, Prospective Clinical Trial Comparing the Impact of Legumes vs Corn-soy Flour on Environmental Enteric Dysfunction and Stunting in Rural Malawian Children 1-3 Year Olds
Brief Title: The Impact of Legumes vs Corn-soy Flour on Environmental Enteric Dysfunction in Rural Malawian Children 1-3 Year Olds
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: LG2
Record Dates: First submitted 2015-06-09; First posted 2015-06-15 (Estimated); Last update posted 2017-05-11 (Actual); Status verified 2017-05

CONDITIONS: Environmental Enteropathy

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Cowpeas (Experimental): Cowpea supplementary food that will be approximately 15% of the calculated total daily intake. Children will receive the food for 12 months.
  Interventions: Dietary Supplement: cowpeas complementary food
- Common bean (Experimental): Common bean supplementary food that will be approximately 15% of the calculated total daily intake. Children will receive the food for 12 months.
  Interventions: Dietary Supplement: common bean complementary food
- Corn Soy Flour (Active Comparator): Corn flour with 10% soy supplementary food that will be approximately 15% of the calculated total daily intake. Children will receive the food for 12 months.
  Interventions: Dietary Supplement: corn-soy flour

INTERVENTIONS:
Dietary Supplement: cowpeas complementary food — cowpeas supplementary food that will be approximately 15% of the calculated total daily intake. Children will receive the food for 12 months.
  Arms: Cowpeas
Dietary Supplement: corn-soy flour — Corn-soy flour supplementary food that will be approximately 15% of the calculated total daily intake. Children will receive the food for 12 months.
  Arms: Corn Soy Flour
Dietary Supplement: common bean complementary food — common bean supplementary food that will be approximately 15% of the calculated total daily intake. Children will receive the food for 12 months.
  Arms: Common bean

SUMMARY:
To determine if 12 months of legume-based complementary foods is effective in reducing or reversing EED and linear growth faltering in a cohort of Malawian children, aged 12-35 months to see if these improvements are correlated with specific changes in the enteric microbiome.

ELIGIBILITY:
Inclusion Criteria:

* children residing in catchment area of Limela, Machinga District and N tenda (Chikwawa District), Malawi
* aged 12-35 months
* youngest eligible child in each household

Exclusion Criteria:Unable to drink 20 mL of sugar water

* Demonstrating evidence of severe acute malnutrition, WHZ < or = -3, presence of bi-pedal pitting edema
* Apparent need for acute medical treatment for an illness or injury
* Caregiver refusal to participate and return for 3, 6 and 12 month follow-ups

Ages: 12 Months to 35 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 337 (Actual)
Dates: Start 2015-08 (Actual); Primary Completion 2016-12 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Dual Sugar Absorption Test | 3 months
  lactulose-mannitol ratio in urine
Dual Sugar Absorption Test | 6 months
  lactulose-mannitol ratio in urine
Dual Sugar Absorption Test | 12 months
  lactulose-mannitol ratio in urine

SECONDARY OUTCOMES:
Lactulose Excretion | 3 months
  percentage of ingested lactulose excreted in urine
Lactulose Excretion | 6 months
  percentage of ingested lactulose excreted in urine
Lactulose Excretion | 12 months
  percentage of ingested lactulose excreted in urine
Mannitol Excretion | 3 months
  percentage of ingested mannitol excreted in urine
Mannitol Excretion | 6 months
  percentage of ingested mannitol excreted in urine
Mannitol Excretion | 12 months
  percentage of ingested mannitol excreted in urine

CONTACTS AND LOCATIONS:
Overall Officials: Mark Manary, MD, Principal Investigator — Washington University School of Medince
Locations (1):
- Blantyre, Malawi

REFERENCES:
- [Derived] Kaimila Y, Pitman RT, Divala O, Hendrixson DT, Stephenson KB, Agapova S, Trehan I, Maleta K, Manary MJ. Development of Acute Malnutrition Despite Nutritional Supplementation in Malawi. J Pediatr Gastroenterol Nutr. 2019 May;68(5):734-737. doi: 10.1097/MPG.0000000000002241. PMID 31022095
- [Derived] Borresen EC, Zhang L, Trehan I, Nealon NJ, Maleta KM, Manary MJ, Ryan EP. The Nutrient and Metabolite Profile of 3 Complementary Legume Foods with Potential to Improve Gut Health in Rural Malawian Children. Curr Dev Nutr. 2017 Sep 21;1(10):e001610. doi: 10.3945/cdn.117.001610. eCollection 2017 Oct. PMID 29955682
- [Derived] Agapova SE, Stephenson KB, Divala O, Kaimila Y, Maleta KM, Thakwalakwa C, Ordiz MI, Trehan I, Manary MJ. Additional Common Bean in the Diet of Malawian Children Does Not Affect Linear Growth, but Reduces Intestinal Permeability. J Nutr. 2018 Feb 1;148(2):267-274. doi: 10.1093/jn/nxx013. PMID 29490090
- [Derived] Trehan I, Benzoni NS, Wang AZ, Bollinger LB, Ngoma TN, Chimimba UK, Stephenson KB, Agapova SE, Maleta KM, Manary MJ. Common beans and cowpeas as complementary foods to reduce environmental enteric dysfunction and stunting in Malawian children: study protocol for two randomized controlled trials. Trials. 2015 Nov 14;16:520. doi: 10.1186/s13063-015-1027-0. PMID 26578308